CLINICAL TRIAL: NCT00534430
Title: Phase II Study of IV Busulfan Combined With 12 cGy of Fractionated Total Body Irradiation (FTBI) and Etoposide (VP-16) as a Preparative Regimen for Allogeneic Bone Marrow Transplantation for Patients With Advanced Hematological Malignancies
Brief Title: Busulfan, Etoposide, and Total-Body Irradiation in Treating Patients Undergoing Donor Stem Cell or Bone Marrow Transplant for Advanced Hematologic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99041; P30CA033572 (NIH); CHNMC-99041; CDR0000564777 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Results first posted 2023-10-10 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; adult acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; blastic phase chronic myelogenous leukemia; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Congenital Abnormalities; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis; Anemia, Refractory, with Excess of Blasts | interventions — Busulfan; Cyclosporine; Etoposide; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

ARMS (1):
- Busulfan, FTBI and VP16 (Experimental): IV Busulfan + 12 cGy FTBI + VP16 prior to allogeneic Bone Marrow Transplant
  Interventions: Drug: busulfan; Drug: cyclosporine; Drug: etoposide; Drug: mycophenolate mofetil; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: total-body irradiation

INTERVENTIONS:
Drug: busulfan
Drug: cyclosporine
Drug: etoposide
Drug: mycophenolate mofetil
Procedure: allogeneic bone marrow transplantation
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: total-body irradiation

SUMMARY:
RATIONALE: Giving chemotherapy and total-body irradiation before a donor stem cell transplant or a donor bone marrow transplant helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving mycophenolate mofetil and cyclosporine before and after transplant may stop this from happening.

PURPOSE: This phase II trial is studying the side effects and best way to give busulfan together with etoposide and total-body irradiation and to see how well they work in treating patients who are undergoing a donor stem cell or bone marrow transplant for advanced hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the efficacy of a preparative regimen comprising dose targeted busulfan, etoposide, and fractionated total-body irradiation followed by allogeneic hematopoietic stem cell or bone marrow transplantation in patients with advanced hematologic malignancies.
* To determine the efficacy of this regimen in patients with acute myeloid leukemia in first remission with unfavorable cytogenetics.
* To evaluate the early and late toxicities of this regimen.

OUTLINE:

* Preparative chemotherapy regimen: Patients receive busulfan IV over 2 hours once every 6 hours on days -14 to -8 for a total of 16 doses and etoposide IV on day -3.* NOTE: *Patients also receive oral or IV dilantin 1-3 times daily on days -18 to -5 for prophylaxis of grand mal seizures.
* Fractionated total-body irradiation (FTBI): Patients undergo FTBI on days -7 to -4 for a total of 10 fractions.
* Allogeneic transplantation: Patients undergo allogeneic peripheral blood stem cell transplantation or bone marrow transplantation on day 0.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive cyclosporine IV or orally on days -1 to 50 followed by a taper to day 180 in the absence of GVHD. Patients also receive mycophenolate mofetil orally or IV over 2 hours twice daily on days 0-27, followed by a taper until day 56.

After completion of study treatment, patients are followed annually for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Acute myeloid leukemia (AML)

    * Failed remission induction therapy or in relapse beyond second remission
    * In first remission with poor risk cytogenetics (e.g., 11q abnormalities, -7, -5, complex abnormalities [i.e., > 3 abnormalities, 6;9 translocation and 3q abnormalities del (7q), del (5q), complex abnormalities ≥ abnormalities, 9q, 20q, 21q, 17q, t(9;21)])
  * Acute lymphoblastic leukemia (ALL)

    * Failed remission induction therapy or in relapse beyond second remission
  * Blastic phase chronic myelogenous leukemia
  * Refractory anemia with excess blasts
  * Refractory anemia with excess blasts in transformation
* HLA -A, -B, -C, -DR identical sibling donor match available
* No relapse after prior bone marrow transplantation

PATIENT CHARACTERISTICS:

* Cardiac ejection fraction ≥ 50%
* Serum creatinine ≤ 1.2 times upper limit of normal (ULN) or creatinine clearance > 80 mL/min
* Bilirubin ≤ 1.5 times ULN
* AST and ALT < 5 times ULN
* FEV_1 ≥ 50% of predicted normal
* DLCO ≥ 50% of predicted normal
* No psychological or medical condition that would preclude allogeneic transplantation (in the opinion of the treating physician)
* Not pregnant
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 28 days since prior induction or reinduction therapy
* Prior etoposide and busulfan allowed
* No prior radiation therapy that would exclude total-body irradiation

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2000-02-29 (Actual); Primary Completion 2010-04-12 (Actual); Study Completion 2026-03-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony S. Stein, MD, Study Chair — City of Hope Comprehensive Cancer Center

RESULTS

PARTICIPANT FLOW:
Groups:
- Busulfan, Fractionated Total Body Irradiation (FTBI) + Etoposide (VP16): IV Busulfan + 12 cGy Fractionated Total Body Irradiation (FTBI) + Etoposide (VP16) prior to allogeneic Bone Marrow Transplant
  busulfan
  cyclosporine
  etoposide
  mycophenolate mofetil
  allogeneic bone marrow transplantation
  allogeneic hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
  total-body irradiation
Period: Overall Study
Arm/Group | Busulfan, Fractionated Total Body Irradiation (FTBI) + Etoposide (VP16)
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Enrolled on protocol after screening for eligiblility
Groups:
- Busulfan, FTBI and VP16: IV Busulfan + 12 cGy FTBI + VP16 prior to allogeneic Bone Marrow Transplant
  busulfan
  cyclosporine
  etoposide
  mycophenolate mofetil
  allogeneic bone marrow transplantation
  allogeneic hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
  total-body irradiation
Arm/Group | Busulfan, FTBI and VP16
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 37 [19 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6
  Hispanic | 2
  White, Not Hispanic | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
Patient Assessment of Mortality (PAM) Score [Median (Full Range); unit: units on a scale] — A risk score for mortality after allogeneic hematopoietic cell transplantation. Ann Intern Med 2006; 144(6):407-414. Parimon T, Au DH, Martin PH, Chien JW. "We generated 4 categories of PAM scores by setting cutoffs according to the probability of death. Scores ranged from 9 to 16 for category 1 (probability of death, < 25%), from 17 to 23 for category 2 (probability of death, 25% to 50%), from 24 to 30 for category 3 (probability of death, 50% to 75%), and from 31 to 44 for category 4 (probability of death, > 75%)."
  units on a scale | 26 [22 to 34]
Disease Status at Transplant [Count of Participants; unit: Participants] — Disease classification was based on WHO criteria [Vardiman, Blood 2002]: Acute myeloid leukemia (AML), Acute lymphoblastic leukemia (ALL), and untreated refractory anemia with excess blasts in transformation (RAEB-t).
  Participants
    AML in First Complete Remission | 6
    AML in First Relapse | 6
    AML in Induction Failure | 10
    untreated RAEB-t | 2
    ALL in First Relapse | 1
    ALL in Second Relapse | 1
    ALL in Induction Failure | 4
Cytogenetics [Count of Participants; unit: Participants] — Cytogenetics were based on Southwest Oncology Group criteria [Leith CP, Blood 1997; Pullarkat V, Blood 2008].
  Intermediate: normal and all other cytogenetic abnormalities. Unfavorable: -5/5q-, -7/7q-, inv(3), 11q abn, 17p abn or i(17q), del(20q), dmins/hsrs, +13, t(9; 22), complex (>3 abn) karyotypes.
  Indeterminate: all other clonal cytogenetic abnormalities.
  Participants
    Indeterminate | 1
    Intermediate | 14
    Unfavorable | 15
Stem Cell Source [Count of Participants; unit: Participants]
  Bone Marrow | 1
  Peripheral Blood | 29
WBC pre-conditioning [Median (Full Range); unit: x10^9 cells/L] — Population: Patients with active disease
  x10^9 cells/L
    number analyzed (Participants) | 24
    (all) | 3.4 [0.9 to 29.2]
Percent Blasts in Bone Marrow [Median (Full Range); unit: percent of leukocytes] — Population: Patients with active disease
  percent of leukocytes
    number analyzed (Participants) | 24
    (all) | 16.5 [0 to 95]
Percent Blasts in Peripheral Blood [Median (Full Range); unit: percent of leukocytes] — Population: Patients with Active Disease
  percent of leukocytes
    number analyzed (Participants) | 24
    (all) | 3.5 [0 to 92]

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 5 Years Post-Transplant.
Description: Kaplan-Meier estimate of an event of death estimated at five years post-transplant. 95% confidence intervals were calculated from the logit transform of the Greenwood variance. The transformation was necessary to keep the estimate within the probability space of 0 to 100%.
Time Frame: Date of Transplant to Five Years post-Transplant
Population: The Full Study Population
Measure: Number (95% Confidence Interval); unit: percentage of survival probability
Arm/Group | Busulfan, FTBI and VP16
Number analyzed (Participants) | 30
percentage of survival probability | 40 [23 to 57]

2. Primary Outcome: Disease-free Survival at Five Years Post-transplant
Description: Kaplan-Meier estimate of an event of relapse or death estimated at five years post-transplant. 95% confidence intervals were calculated from the logit transform of the Greenwood variance. The transformation was necessary to keep the estimate within the probability space of 0 to 100%.
Time Frame: Date of transplant to five years post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of survival probability
Arm/Group | Busulfan, FTBI and VP16
Number analyzed (Participants) | 30
percentage of survival probability | 40 [23 to 57]

3. Primary Outcome: Overall Survival Comparing Diagnosis Groups
Description: as for outcome 1
Time Frame: Date of Transplant to Five Years post-Transplant
Population: Study cohort separated into four disease groups.
Measure: Number (95% Confidence Interval); unit: percentage of survival probability
Groups:
- AML/1CR: Acute Myelogenous Leukemia Transplanted in First Complete Remission
- AML/R1: Acute Myelogenous Leukemia Transplanted in First Relapse
- AML/IF: Acute Myelogenous Leukemia Transplanted in Induction Failure
- Active ALL: Active Acute Lymphocytic Leukemia
Arm/Group | AML/1CR | AML/R1 | AML/IF | Active ALL
Number analyzed (Participants) | 6 | 6 | 10 | 6
percentage of survival probability | 67 [20 to 90] | 50 [11 to 80] | 30 [7 to 38] | 33 [5 to 38]
Statistical Analysis 1: Comparison: AML/1CR vs AML/R1 vs AML/IF vs Active ALL; Log-rank test. (Mantel-Haenszel test). Null hypothesis is all four groups are statistically from the same population. Alternative hypothesis is that at least one of the groups is from a population different from the remaining groups. Anticipated sample-sizes comparing Active ALL (anticipated N= 12) with the combined AML patients (anticipated N=38) was deemed to be too small for formal hypothesis testing; Test type: Equivalence — Given the small sample-size of the disease sub-groups, this was a hypothesis generating study; p > 0.05, Log Rank — Not adjusted for multiple comparisons. A-priori threshold for statistical significance was 0.05; No adjustments; Median Difference (Net) = 0

4. Primary Outcome: Cumulative Incidence of Relapse With Transplant-related Death as the Competing Risk: Diagnosis Groups Are Compared.
Description: Fine and Gray estimate of cumulative incidence of Relapse, with Death as the competing risk. Estimate is at five years post-transplant. Ninety-five percent confidence interval is by logit transformation of Greenwood variance to keep the interval within the probability space of 0% to 100%.
Time Frame: Date of Transplant to Five Years post-Transplant. Estimate is at Five Years post-Transplant.
Measure: Number (95% Confidence Interval); unit: percentage of relapse probability
Arm/Group | AML/1CR | AML/R1 | AML/IF | Active ALL
Number analyzed (Participants) | 6 | 6 | 10 | 6
percentage of relapse probability | 0 [0 to 0] | 0 [0 to 0] | 30 [9 to 65] | 50 [13 to 87]
Statistical Analysis 1: Comparison: AML/1CR vs AML/R1 vs AML/IF vs Active ALL; Gray's estimate. (Fine and Gray). Null hypothesis is all four groups are statistically from the same population. Alternative hypothesis is that at least one of the groups is from a population different from the remaining groups. Anticipated sample-sizes comparing Active ALL (anticipated N= 12) with the combined AML patients (anticipated N=38) was deemed to be too small for formal hypothesis testing; Test type: Equivalence — Given the small sample-size of the disease sub-groups, this was a hypothesis generating study; p > 0.05, Gray's Test — Not adjusted for multiple comparisons. A-priori threshold for statistical significance was 0.05; No adjustments; Median Difference (Net) = 0

ADVERSE EVENTS:
Time Frame: From the start time of the study treatment up to Day 100 post-transplant
Description: Systematic Assessment: See the time periods, above.
Arm/Group | Busulfan, FTBI and VP16
All-Cause Mortality (participants affected / at risk) | 18/30
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Busulfan, FTBI and VP16 (N=30)
Leukocytes (total WBC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Busulfan, FTBI and VP16 (N=30)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 3
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 3
Allergy/Immunology - Other: DRY NOSE (Immune system disorders) | 1
Allergy/Immunology - Other: ENGRAFTMENT SYNDROME (Immune system disorders) | 1
Auditory/Ear - Other: DECREASED HEARING DUETO MEDS (AZITHROMYCIN) (Ear and labyrinth disorders) | 1
Auditory/Ear - Other: PLUGGED EARS (Ear and labyrinth disorders) | 1
Otitis, external ear (non-infectious) (Ear and labyrinth disorders) | 1
Graft versus host disease (General disorders) | 14
Veno-Occlusive Disease (VOD) (General disorders) | 3
Blood/Bone Marrow - Other (Specify, __) (Blood and lymphatic system disorders) | 1
Bone marrow cellularity (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 24
Hemoglobin for leukemia studies or bone marrow infiltrative/ myelophthisic processes. (Blood and lymphatic system disorders) | 1
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 1
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1
Leukocytes (total WBC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 23
Lymphopenia (Blood and lymphatic system disorders) | 22
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 24
Platelets (Blood and lymphatic system disorders) | 1
Platelets for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 25
Transfusion: Platelets (Blood and lymphatic system disorders) | 1
Transfusion: Platelets for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 23
Transfusion: pRBCs (Blood and lymphatic system disorders) | 2
Transfusion: pRBCs for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 25
Acute graft versus host disease (GVHD) (COH) (General disorders) | 15
Chronic graft versus host disease (GVHD) (COH) (General disorders) | 1
Cardiac Arrhythmia - Other (Specify, __) (Cardiac disorders) | 1
Supraventricular and nodal arrhythmia (Cardiac disorders) | 19
Ventricular arrhythmia (Cardiac disorders) | 1
Cardiac General - Other (Specify, __) (Cardiac disorders) | 1
Cardiac General - Other: CARDIOMEGALY (Cardiac disorders) | 2
Hypertension (Cardiac disorders) | 17
Hypotension (Cardiac disorders) | 8
Myocarditis (Cardiac disorders) | 1
Edema (Vascular disorders) | 20
INR (International Normalized Ratio of prothrombin time) (Vascular disorders) | 8
PTT (Partial Thromboplastin Time) (Vascular disorders) | 4
Constitutional Symptoms - Other (Specify, __) (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 23
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 12
Insomnia (General disorders) | 13
Rigors/chills (General disorders) | 20
Sweating (diaphoresis) (General disorders) | 3
Weight gain (General disorders) | 4
Weight gain - Veno-Occlusive Disease (VOD) for BMT studies if specified in the protocol. (General disorders) | 2
Weight loss (General disorders) | 16
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: ACTINIC PARAKERATIONS (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: BRUISE ON RIGHT ARM (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: BURNING SENSATION IN ARM PITS (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: CONTACT DERMATITIS (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: DIFFUSE ERYTHEMATOUS SCROTUM (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: EDEMA DUE TO BM BIOPSY (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: FACIAL PLETHORA (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: FACIAL SWELLING (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: INGROWN TOENAIL (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: INTRAVASCULAR MICROTHROMBI - LEFT THIGH (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: LEFT HIP ABRASION (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: LIP LESION (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: PALLOR (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: PAROTID SWELLING (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: PERI-RECTAL EXCORIATION (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: PERIANAL AREA SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: PERIRECTAL AREA SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: PERIRECTAL ULCER (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: RASH SECONDARY CHEMO (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: REDNESS ON SCROTUM (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: ROSACEA (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: SCROTAL RASH (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: SKIN/JAUNDICE (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: UP ORAL ULCER (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: VP-16 RASH (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: VP-16 SKIN RASH (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 7
Flushing (Skin and subcutaneous tissue disorders) | 8
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 10
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 5
Nail changes (Skin and subcutaneous tissue disorders) | 2
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 12
Pruritus/itching (Skin and subcutaneous tissue disorders) | 9
Rash/dermatitis associated with high-dose chemotherapy or BMT studies. (Skin and subcutaneous tissue disorders) | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7
Rash/desquamation associated with graft versus host disease (GVHD). (Skin and subcutaneous tissue disorders) | 18
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 10
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 1
Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 6
Anorexia (Gastrointestinal disorders) | 25
Ascites (non-malignant) (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 7
Dehydration (Gastrointestinal disorders) | 12
Diarrhea (Gastrointestinal disorders) | 11
Diarrhea associated with graft versus host disease (GVHD) (Gastrointestinal disorders) | 14
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 4
Dysphagia-esophageal related to radiation (Gastrointestinal disorders) | 2
Esophagitis (Gastrointestinal disorders) | 9
Flatulence (Gastrointestinal disorders) | 1
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 2
Gastrointestinal - Other: ABDOMINAL BLOATING (Gastrointestinal disorders) | 1
Gastrointestinal - Other: ABDOMINAL BLOATNESS (Gastrointestinal disorders) | 1
Gastrointestinal - Other: ABDOMINAL CRAMPS (Gastrointestinal disorders) | 1
Gastrointestinal - Other: ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1
Gastrointestinal - Other: CHOLECYSTITIS (Gastrointestinal disorders) | 1
Gastrointestinal - Other: DRY HEAVES (Gastrointestinal disorders) | 4
Gastrointestinal - Other: DRY MOUTH (Gastrointestinal disorders) | 1
Gastrointestinal - Other: EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 1
Gastrointestinal - Other: ERYTHEMA STOMACH (Gastrointestinal disorders) | 1
Gastrointestinal - Other: ESOPHAGEAL DISCOMFORT (Gastrointestinal disorders) | 1
Gastrointestinal - Other: FREQUENT STOOLS (NOT DIARRHEA) (Gastrointestinal disorders) | 1
Gastrointestinal - Other: GAGGING (Gastrointestinal disorders) | 1
Gastrointestinal - Other: GERD (Gastrointestinal disorders) | 1
Gastrointestinal - Other: GURGLY STOMACH (Gastrointestinal disorders) | 1
Gastrointestinal - Other: INCREASED SALIVATION (Gastrointestinal disorders) | 1
Gastrointestinal - Other: ORAL THRUSH (Gastrointestinal disorders) | 1
Gastrointestinal - Other: RECTAL LESION (Gastrointestinal disorders) | 1
Gastrointestinal - Other: RED THROAT (Gastrointestinal disorders) | 1
Gastrointestinal - Other: RETCHING (Gastrointestinal disorders) | 2
Gastrointestinal - Other: SCRATCHY THROAT (Gastrointestinal disorders) | 1
Gastrointestinal - Other: SMALL POLYPS STOMACH (Gastrointestinal disorders) | 1
Gastrointestinal - Other: SWELLING OF CHECKS (Gastrointestinal disorders) | 1
Gastrointestinal - Other: UPPER GI/GVHD (Gastrointestinal disorders) | 1
Gastrointestinal - Other: WRECHING (Gastrointestinal disorders) | 1
Gastrointestinal - Other: WRETCHING (Gastrointestinal disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 16
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 2
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 25
Salivary gland changes/saliva (Gastrointestinal disorders) | 5
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT studies, if specified in the protocol. (Gastrointestinal disorders) | 24
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 22
Hematemesis (Vascular disorders) | 8
Hematuria (in the absence of vaginal bleeding) (Vascular disorders) | 3
Hemoptysis (Vascular disorders) | 3
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Vascular disorders) | 16
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Vascular disorders) | 14
Melena/GI bleeding (Vascular disorders) | 2
Rectal bleeding/hematochezia (Vascular disorders) | 5
Hemorrhage, GU (Vascular disorders) | 9
Hemorrhage, pulmonary/upper respiratory (Vascular disorders) | 9
Hemorrhage/Bleeding - Other: BLEEDING FROM PENIS MEATUS (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: BLEEDING FROM SCRATCH (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: BLOOD IN SPUTUM (Vascular disorders) | 2
Hemorrhage/Bleeding - Other: BLOOD TINGLED MUCUS (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: HEMORRHOIDS (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: SPUTUM WITH BLOODSTREAM (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: SUBCONJUNCTIVAL HEMORRHAGE (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: TELANGIECTASIA CHEST (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: TONGUE BLEEDING (Vascular disorders) | 1
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Vascular disorders) | 8
Bilirubin associated with graft versus host disease (GVHD). (Hepatobiliary disorders) | 3
Hepatic enlargement (Hepatobiliary disorders) | 2
Hepatobiliary/Pancreas - Other: JAUNDICE (Hepatobiliary disorders) | 1
Febrile neutropenia (fever of unknown origin) (Infections and infestations) | 22
Infection - Other (Specify, __) (Infections and infestations) | 1
Infection - Other: ORAL CANDIDIASIS (Infections and infestations) | 1
Infection - Other: UPPER RESPIRATORY INFECTION (Infections and infestations) | 1
Infection with unknown ANC (Infections and infestations) | 11
Infection (documented) with grade 3 or 4 neutropenia (Infections and infestations) | 10
Infection with unknown ANC (Infections and infestations) | 1
Infection without neutropenia (Infections and infestations) | 21
Infection, Bacterial (COH) (Infections and infestations) | 20
Infection, Fungal (COH) (Infections and infestations) | 9
Infection, Viral (Infections and infestations) | 18
Lymphatics - Other: LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1
Lymphatics CERVICAL LYMPHOADENOPATHY (Blood and lymphatic system disorders) | 1
Lymphatics MILD LYMPHEDEMIA (NECK) (Blood and lymphatic system disorders) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 26
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 24
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 2
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 26
Alkaline phosphatase (Metabolism and nutrition disorders) | 18
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 2
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 21
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 16
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 4
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 25
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 12
Creatinine (Metabolism and nutrition disorders) | 24
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 26
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 4
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 10
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 27
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 16
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 14
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 27
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 4
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 27
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 11
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal/Soft Tissue - Other: DEGERATIVE CHANGES IN ANTERIOR THORACIC SPINE (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue - Other: HAND CRAMPS (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue - Other: MUSCLE CRAMPS (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal/Soft Tissue - Other: MUSCLE CRAMPS-FINGERS (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue - Other: MUSCLE SPANAM (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue - Other: MUSCLE SPASM (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue - Other: NUMBNESS, TINGLING (Musculoskeletal and connective tissue disorders) | 1
Ataxia (incoordination) (Nervous system disorders) | 2
Confusion (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 11
Hallucinations (Nervous system disorders) | 5
Mood alteration (Nervous system disorders) | 15
Neurology - Other: ADJUSTMENT DISORDER WITH MIXED ANXIETY AND DEPRESSION (Nervous system disorders) | 1
Neurology - Other: METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1
Neurology - Other: NIGHTMARES (Nervous system disorders) | 1
Neurology - Other: PANIC ATTACK (Nervous system disorders) | 1
Neuropathy: motor (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 3
Personality/behavioral (Nervous system disorders) | 1
Psychosis (hallucinations/delusions) (Nervous system disorders) | 1
Pyramidal tract dysfunction (increased tone, hyperreflexia, pos Babinski, decreased motor coord (Nervous system disorders) | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 7
Syncope (fainting) (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 9
Dry eye syndrome (Eye disorders) | 6
Ocular surface disease (Eye disorders) | 5
Ocular/Visual - Other: CHEMON'S--SCLERAL EDEMA (Eye disorders) | 1
Ocular/Visual - Other: ICTERIC SCLERAE (Eye disorders) | 1
Ocular/Visual - Other: JAUNDICED SCLERAL (Eye disorders) | 1
Ocular/Visual - Other: RED EYES (Eye disorders) | 1
Ocular/Visual - Other: REDNESS (NOT DRY) (Eye disorders) | 1
Ocular/Visual - Other: YELLOW DISCHARGE FROM THE EYES (Eye disorders) | 1
Vision-blurred vision (Eye disorders) | 1
Pain (General disorders) | 23
Pain - Other: ARM PIT PAIN (General disorders) | 1
Pain - Other: BACK PAIN (General disorders) | 2
Pain - Other: BODY ACHE (General disorders) | 1
Pain - Other: CATHETER PAIN (General disorders) | 1
Pain - Other: CRAMPING (ABDOMINAL) (General disorders) | 1
Pain - Other: DRY HEAVES (General disorders) | 1
Pain - Other: EAR PAIN (General disorders) | 1
Pain - Other: EPIGASTRIC PAIN (General disorders) | 4
Pain - Other: GENERALIZED BODY PAIN (General disorders) | 2
Pain - Other: HANDS PAIN (General disorders) | 1
Pain - Other: HICKMAN CATHETER PAIN (General disorders) | 1
Pain - Other: HICKMAN SITE PAIN (General disorders) | 2
Pain - Other: HIP PAIN (DUE TO BIOPSY) (General disorders) | 1
Pain - Other: INGROWN TOENAIL PAIN (General disorders) | 1
Pain - Other: KNEE PAIN (General disorders) | 1
Pain - Other: LEG PAIN (General disorders) | 1
Pain - Other: LOW BACK PAIN (General disorders) | 1
Pain - Other: MOUTH PAIN (General disorders) | 3
Pain - Other: NECK PAIN (General disorders) | 2
Pain - Other: PAIN AT RAC SITE (General disorders) | 1
Pain - Other: PAIN FROM BM BIOPSY SITE (General disorders) | 1
Pain - Other: PAIN IN MANDIBLE (General disorders) | 1
Pain - Other: PAIN SYNDROME DUE TO MUCOSITIS (General disorders) | 1
Pain - Other: PAIN TO LYMPH NODE (General disorders) | 1
Pain - Other: PAROTID PAIN (General disorders) | 2
Pain - Other: PERIRECTAL PAIN (General disorders) | 1
Pain - Other: R. ARM PAIN FROM THE FALL (General disorders) | 1
Pain - Other: RAC SITE PAIN (General disorders) | 3
Pain - Other: RIB PAIN (General disorders) | 1
Pain - Other: SCROTAL PAIN (General disorders) | 1
Pain - Other: SHOULDER PAIN (General disorders) | 1
Pain - Other: SKIN PAIN (General disorders) | 1
Pain - Other: SUBMANDIBULAR TENDERNESS (General disorders) | 1
Pain - Other: TENDER PAROTID GLANDS (General disorders) | 1
Pain - Other: THIGH PAIN (General disorders) | 1
Pain - Other: THROAT PAIN (General disorders) | 4
Pain - Other: THROAT PAIN (POSSIBLE URI) (General disorders) | 1
Pain - Other: TONGUE PAIN (General disorders) | 1
Pain - Other: TWINGES FEET (General disorders) | 1
Pain RECTAL PAIN (General disorders) | 1
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 17
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 8
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: DECREASED BREATH SOUND AT LUNG BASES (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: EXCORIATION OF POSTERIOR (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: MILD ELEVATION OF RIGHT HEMIDIAPHRAGM (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary/Upper Respiratory - Other: NASAL STUFFINESS (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory - Other: NASAL/SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: PULMONARY VASCULAR CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: RUNNING NOSE (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: SINUS CONGESTION/RUNNY NOSE (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: SINUS/NOSE CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: TACHYPNEA (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: UPPER AIRWAY OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: URI (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 9
Bladder spasms (Renal and urinary disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 1
Renal/Genitourinary - Other: VAG. DISCHARGE (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1
Libido (Reproductive system and breast disorders) | 1
Vaginitis (not due to infection) (Reproductive system and breast disorders) | 3
Syndromes - Other: RASH GVHD (General disorders) | 1
Tumor lysis syndrome (General disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2004-04-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT00534430/Prot_SAP_000.pdf